CLINICAL TRIAL: NCT00408187
Title: A Phase III, Randomized, Multicentre, Double-Blind, Placebo and Ciclosporin Controlled Study of ISA247 in Plaque Psoriasis Patients
Brief Title: Randomized, Placebo and Ciclosporin Controlled Study of ISA247 in Plaque Psoriasis Patients
Acronym: ESSENCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aurinia Pharmaceuticals Inc. (Industry)
Responsible Party: Robert Huizinga, Isotechnika
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISA05-25
Record Dates: First submitted 2006-12-04; First posted 2006-12-06 (Estimated); Last update posted 2009-07-30 (Estimated); Status verified 2009-07

CONDITIONS: Psoriasis
Keywords: Randomized Controlled Trials; Immunosuppression; Adult; Chronic Disease; Dermatologic Agents; Female; Humans; Male; Middle Aged; Severity of Illness Index; Treatment Outcome; Quality of Life; Double-Blind Method
MeSH Terms: conditions — Psoriasis; Chronic Disease | interventions — voclosporin; Cyclosporine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1. (Active Comparator)
  Interventions: Drug: voclosporin
- 3. (Placebo Comparator)
  Interventions: Drug: Placebo
- 2. (Active Comparator)
  Interventions: Drug: Ciclosporin

INTERVENTIONS:
Drug: voclosporin — voclosporin 0.4 mg/kg po BID
  Arms: 1.
Drug: Ciclosporin — ciclosporin 1.5 mg/kg po BID
  Arms: 2.
Drug: Placebo — Placebo
  Arms: 3.

SUMMARY:
The purpose of this study is to determine the safety and efficacy of voclosporin in patients with plaque psoriasis.

DETAILED DESCRIPTION:
Psoriasis is a chronic skin condition that can have a significant impact on a patient's physical and mental well being. The most common form of psoriasis is plaque psoriasis. Targeted treatments in psoriasis have been reported recently, yet ciclosporin, a calcineurin inhibitor (CNi) remains one of the treatments which has the greatest efficacy. Voclosporin represents the possibility of a calcineurin inhibitor which is not only as efficacious as ciclosporin A, but also has an improved toxicity profile.

ELIGIBILITY:
Inclusion Criteria:

* Aged greater than or equal to 18 years of age inclusive at time of screening.
* Diagnosed with plaque psoriasis greater than or equal to 6 months prior to screening.
* Diagnosis of stable, plaque psoriasis; i.e. psoriasis must not be spontaneously improving or worsening in the 4 weeks prior to the screening visit.
* Psoriasis failing at least one systemic treatment regimen or where other systemic therapies are contraindicated or where tolerability is an issue.
* Plaque psoriasis involving greater than or equal to 10% of the body surface area and a SPGA score greater than or equal to 3 at screening and prior to randomization at the day 0 visit.
* Not pregnant or nursing.
* Sexually active women of childbearing potential or less than 1 year post-menopausal and sexually active men who are not surgically sterile must use a reliable form of birth control during study treatment and for at least 3 months after the last dose of study drug. Surgically sterile females are not considered to be of childbearing potential. Reliable forms of birth control include oral or depot contraceptives, and double-barrier methods.
* Written informed consent prior to washout and screening procedures.
* Able to keep study appointments and cooperate with all study requirements, in the opinion of the Investigator.

Exclusion Criteria:

* Has generalized erythrodermic, guttate, or pustular psoriasis.
* Have other dermatoses that would interfere with the evaluation of psoriasis, at the discretion of the Investigator.
* A current malignancy or history of malignancy within 5 years or a history of lymphoma at any time. Subjects can be enrolled with a history of squamous or basal cell carcinoma that has been surgically excised or removed with curettage and electrodesiccation.
* Has a current, uncontrolled bacterial, viral, or fungal infection that requires intravenous antibiotics or antifungals or has had such infections within 60 days prior to screening.
* A known history of tuberculosis.
* Serologic evidence or known latent HIV, HBV or HCV virus.
* Uncontrolled hypertension of systolic blood pressure greater than or equal to 160 mmHg or diastolic blood pressure greater than or equal to 90 mmHg.
* MDRD GFR < 60 mL/min.
* Variation between the screening and Visit 1 SCr greater than or equal to 30%.
* ALT, AST, GGT greater than or equal to 2x upper limit of normal (ULN).
* White blood cell count less than or equal to 2.8 x 10 to the ninth power/L.
* Requires the following prohibited medications or treatments during the washout or treatment period: drugs potentiating the nephrotoxicity of voclosporin, drugs interfering with its pharmacokinetics, drugs considered to contribute to psoriasis flare; or, systemic and topical psoriasis medication that may interfere with assessment of study drug efficacy.
* Has used any investigational drug or device within 30 days or 10 half lives (whichever is longer) prior to the screening visit.
* Current participation in another clinical trial of any drug or biological agent.
* Has taken biological agent(s), except flu shots, tetanus shots, or boosters, within 3 months of randomization. Biological agents include any virus, live vaccine, therapeutic serum, toxin, antitoxin, monoclonal antibodies or analogous product applicable to the prevention, treatment, or cure of diseases or injuries of man.
* Previous exposure to voclosporin.
* A history of clinically defined allergy to ciclosporin, constituents of Neoral or any of the constituents of the ISA247 formulation.
* A history of alcoholism or drug addiction.
* Weighs < 45kg (99 lbs).
* A history of disease, including mental/emotional disorder that would interfere with the subject's participation in the study, in the evaluation of his/her response or that might cause the administration of voclosporin to pose a significant risk to the subject, in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 642 (Actual)
Dates: Start 2006-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Superiority in the proportion of subjects achieving a score of "clear" or "almost clear" in the Static Physician's Global Assessment (SPGA) score | Twelve weeks of treatment

SECONDARY OUTCOMES:
To show non-inferiority of voclosporin compared to ciclosporin in the proportion of subjects achieving a score of "clear" or "almost clear" in the Static Physician's Global Assessment (SPGA) score at | Twelve weeks of treatment
Superiority in de novo hypertriglyceridemia, defined as proportion of patients developing fasting triglycerides greater than or equal to 1.7 mmol/L | Twenty four weeks of treatment
Superiority in de novo hypertension, defined as proportion of patients developing blood pressure greater than or equal to 140 mmHg (systolic) or greater than or equal to 90 mmHg (diastolic) | Twenty four weeks of treatment
Superiority of renal function, defined as the proportion of patients experiencing a confirmed greater than or equal to 30% rise in serum creatinine | Twenty four weeks of treatment
Superiority in proportion of patients achieving a 75% reduction in the Psoriasis Area and Severity Index (PASI) score (PASI-75) | Twelve weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Gulliver, M.D., Principal Investigator — NewLab Clinical Research; Vincent Ho, M.D., Principal Investigator — UBC; Andrzej Langner, Prof. Dr., Principal Investigator — IWOLANG; Thomas A. Luger, Prof. Dr., Principal Investigator — Universität Münster; Slawomir Majewski, Prof. Dr., Principal Investigator — Akademia Medyczna; Wolfram Sterry, Prof. Dr., Principal Investigator — Charite Universitatsmedizin Berlin
Locations (41):
- Canada (13):
  - Isotechnika Investigational Site, Edmonton, Alberta
  - Isotechnika Investigational Site, Surrey, British Columbia
  - Isotechnika Investigational Site, Vancouver, British Columbia
  - Isotechnika Investigational Site, St. John's, Newfoundland and Labrador
  - Isotechnika Investigational Site, Halifax, Nova Scotia
  - Isotechnika Investigational Site, Barrie, Ontario
  - Isotechnika Investigational Site, London, Ontario
  - Isotechnika Investigational Site, Markham, Ontario
  - Isotechnika Investigational Site, North Bay, Ontario
  - Isotechnika Investigational Site, Ottawa, Ontario
  - Isotechnika Investigational Site, Waterloo, Ontario
  - Isotechnika Investigational Site, Montreal, Quebec
  - Isotechnika Investigational Site, Québec, Quebec
- Germany (16):
  - Isotechnika Investigational Site, Ausburg
  - Isotechnika Investigational Site, Berlin
  - Isotechnika Investigational Site, Bochum
  - Isotechnika Investigational Site, Dresden
  - Isotechnika Investigational Site, Frankfurt
  - Isotechnika Investigational Site, Geiβen
  - Isotechnika Investigational Site, Hamburg
  - Isotechnika Investigational Site, Kiel
  - Isotechnika Investigational Site, Leipzig
  - Isotechnika Investigational Site, Lübeck
  - Isotechnika Investigational Site, Mahlow
  - Isotechnika Investigational Site, Mainz
  - Isotechnika Investigational Site, Münster
  - Isotechnika Investigational Site, Potsdam
  - Isotechnika Investigational Site, Salzwedel
  - Isotechnika Investigational Site, Wuppertal
- Poland (12):
  - Isotechnika Investigational Site, Bialystock
  - Isotechnika Investigational Site, Bydgoszcz
  - Isotechnika Investigational Site, Gliwice
  - Isotechnika Investigational Site, Iwonicz-Zdrój
  - Isotechnika Investigational Site, Krakow
  - Isotechnika Investigational Site, Lodz
  - Isotechnika Investigational Site, Lublin
  - Isotechnika Investigational Site, Poznan
  - Isotechnika Investigational Site, Szczcin
  - Isotechnika Investigational Site, Warsaw
  - Isotechnika Investigational Site, Warzszawa
  - Isotechnika Investigational Site, Zabrze

REFERENCES:
- [Background] Gregory CR, Kyles AE, Bernsteen L, Wagner GS, Tarantal AF, Christe KL, Brignolo L, Spinner A, Griffey SM, Paniagua RT, Hubble RW, Borie DC, Morris RE. Compared with cyclosporine, ISATX247 significantly prolongs renal-allograft survival in a nonhuman primate model. Transplantation. 2004 Sep 15;78(5):681-5. doi: 10.1097/01.tp.0000131950.75697.71. PMID 15371668
- [Background] Stalder M, Birsan T, Hubble RW, Paniagua RT, Morris RE. In vivo evaluation of the novel calcineurin inhibitor ISATX247 in non-human primates. J Heart Lung Transplant. 2003 Dec;22(12):1343-52. doi: 10.1016/s1053-2498(03)00033-0. PMID 14672749
- [Background] Abel MD, Aspeslet LJ, Freitag DG, Naicker S, Trepanier DJ, Kneteman NM, Foster RT, Yatscoff RW. ISATX247: a novel calcineurin inhibitor. J Heart Lung Transplant. 2001 Feb;20(2):161. doi: 10.1016/s1053-2498(00)00290-4. No abstract available. PMID 11250240
- [Background] Bissonnette R, Papp K, Poulin Y, Lauzon G, Aspeslet L, Huizinga R, Mayo P, Foster RT, Yatscoff RW, Maksymowych WP; ISA247 Psoriasis Study Group. A randomized, multicenter, double-blind, placebo-controlled phase 2 trial of ISA247 in patients with chronic plaque psoriasis. J Am Acad Dermatol. 2006 Mar;54(3):472-8. doi: 10.1016/j.jaad.2005.10.061. Epub 2006 Jan 23. PMID 16488299